CLINICAL TRIAL: NCT03401086
Title: Comparison of Kinesiotaping and Pressure Garment on Old Adult Women With Secondary Upper Extremity Lymphedema Following Mastectomy: A Randomized Controlled Trial
Brief Title: Comparison of Kinesiotaping and Pressure Garment on Women With Upper Extremity Lymphedema Following Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahlia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Associate Professor, Ahlia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo University
Record Dates: First submitted 2017-12-25; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The KT group received Kinesio taping application, while the PG group received pressure garment (40-60 mmHg) for at least 15-18 hours per day through the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Kinesio Taping
  Interventions: Other: Kinesio Taping
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Kinesio Taping — Kinesio Taping
  Arms: Study group

SUMMARY:
Breast cancer is a standout amongst the most widely recognized cancer among women. It is observed that upper extremity lymphedema is one of the most dangerous and prevalent complication following breast cancer surgery which prompts functional impairment, psychological disaster and social problems

This study aimed to compare the effects of Kinesio taping and the pressure garment application on secondary lymphedema of the upper extremity and quality of life following mastectomy after breast cancer.

Material and Methods: In this experimental study with pre and post-tests, 66 women with lymphedema following mastectomy were randomly allocated to Kinesio taping (KT) group (n=33) and pressure garment (PG) group (n=33). The KT group received Kinesio taping application, while the PG group received pressure garment (40-60 mmHg) for at least 15-18 hours per day through the study. All patients were evaluated to record the changes of the limb circumference, Shoulder Pain and Disability Index (SPADI), hand grip strength and quality of life at baseline and end of intervention.

DETAILED DESCRIPTION:
66 women with unilateral breast cancer related to lymphedema (stage II and III) for at least for 6 months were invited to participate in the study. Lymphoma was more than 2 cm in arm circumference or less than 8 cm in comparison with the other side. The participants were randomly assigned to 2 groups. Kinesio taping group included 33 patients receiving Kinesio taping (KT) and pressure garment (PG) included 33 patients.

The exclusion criteria were any active disease which leads to swelling, medications, especially diuretics, allergy, infection, pregnancy, heart and kidney diseases, bilateral lymphedema and cellulitis.

All patients were evaluated to record the changes of the limb circumference, Shoulder Pain and Disability Index (SPADI), hand grip strength and quality of life

ELIGIBILITY:
Inclusion Criteria:

* unilateral breast cancer related to lymphedema (stage II and III) for at least for 6 months were invited to participate in the study. Lymphoma was more than 2 cm in arm circumference or less than 8 cm in comparison with the other side.

Exclusion Criteria:

* The exclusion criteria were any active disease which leads to swelling, medications, especially diuretics, allergy, infection, pregnancy, heart and kidney diseases, bilateral lymphedema and cellulitis.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with breast cancer lymphedema after mastetctomy
Enrollment: 66 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Limb circumference | 1 month
  The upper Limbs circumferences were measured by using a tape measure with the patient in prone lying position.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index | 1 month
  Shoulder Pain and Disability Index (SPADI) survey was created to assess the shoulder pain and disability. It incorporates of 13 items that assess two domains: a 5 items that assess pain and an 8 items that evaluate disability.
Hand grip strength | 1 month
  Hand grip strength was evaluated by Dynamometer (78010, Lafayette Instrument Company, Loughboroug, Leics, United Kingdom). The grip strength was measured while the patient was in a standing position with adducted shoulder, flexed elbow 90 degrees and forearm in mid position.
Quality of life | 1 month
  The quality of life was assessed by utilizing cancer-specific questionnaire (EORTC) QLQ-C30 before and after intervention. QLQ-C30 comprised of 30 questions, including functional scores (physical, social, emotional, and cognitive aspects).

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A Tantawy, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Dr Dalia Kamel, Giza
  - Dr Sayed Tanatwy, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tantawy SA, Abdelbasset WK, Nambi G, Kamel DM. Comparative Study Between the Effects of Kinesio Taping and Pressure Garment on Secondary Upper Extremity Lymphedema and Quality of Life Following Mastectomy: A Randomized Controlled Trial. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419847276. doi: 10.1177/1534735419847276. PMID 31068019